CLINICAL TRIAL: NCT01164098
Title: The Use of Rituximab to Prevent Recurrence of Proteinuria in Patients Receiving Kidney Transplant for FSGS
Brief Title: Rituximab to Prevent Recurrence of Proteinuria
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Voluntarily terminated by PI due to lack of feasibility.
Sponsor: George W. Burke (Other)
Collaborators: Genentech, Inc. (Industry); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, George W. Burke, Professor of Surgery, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20100498; 1R01DK090316-01A1 (NIH)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: FSGS; Proteinuria
MeSH Terms: conditions — Proteinuria | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (Active Comparator): Participants will receive Rituximab post within 24 of Kidney Transplant
  Interventions: Drug: Rituximab
- No rituximab (No Intervention): Participants will not receive Rituximab within 24 hours of Kidney Transplant

INTERVENTIONS:
Drug: Rituximab — Induction therapy
  Other Names: Rituxan
  Arms: Rituximab

SUMMARY:
The investigators propose to study novel targets of rituximab in podocytes, with a particular focus on recurrent focal segmental glomerulosclerosis (FSGS). The proposed study has strong clinical implications, since it may extend the approved indications for rituximab treatment to recurrent FSGS as well as to other proteinuric diseases. Furthermore, it will offer new insights into the role of sphyngomyelin related enzymes in podocyte function in health and disease, thus allowing the identification of novel targets for antiproteinuric drug development. Finally, the proposed study offers the opportunity to identify a correlation between the patient's specific clinical outcome and the experimental results obtained after exposing podocytes to patient sera in the presence or absence of rituximab. Therefore, it may lead to the development of an assay for the pre-transplant identification of patients at high-risk for recurrent disease and, among them, may allow the identification of those patients that will respond to rituximab.

DETAILED DESCRIPTION:
A total of 60 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion:

1. Patient has been fully informed and has signed a dated IRB-approval informed consent form.
2. Age 7-65 years.
3. Male and Females diagnosed of FSGS by kidney biopsy. Kidney biopsy report is not required once the physician confirms the diagnosis. Transcribed reports from referring physicians are also valid.

Exclusion:

1. Recipient or donor is seropositive for human immunodeficiency virus (HIV), Hepatitis C viruses, or Hepatitis B virus antigenemia.
2. Patient has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully or carcinoma in situ of the cervix that has been treated successfully.
3. Patient has uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or an active peptic ulcer or any other unstable medical condition that could interfere with study objectives.
4. Patient is pregnant or lactating.
5. Patient has any form of substance abuse, psychiatric disorder or a condition that, in opinion of the investigator, may invalidate communication with the investigator.
6. Patients with a defined genetic cause of FSGS.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessia Fornoni, M.D., Principal Investigator — University of Miami; George W. Burke, M.D., Study Director — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab | No Rituximab
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | No Rituximab | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum of the Urine Protein/Creatinine Ratio Observed Between Post-Transplant Days 3-30.
Description: Primary Outcome - Maximum of the Urine Protein/Creatinine Ratio Observed Between Post-Transplant Days 3-30 will be compared between the two treatment arms using an intent-to-treat approach.
Time Frame: between post-transplant day 3 and day 30
Population: Intent-to-Treat Analysis
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | Rituximab | No Rituximab
Number analyzed (Participants) | 15 | 15
ratio | 1.44 (1.33) | 2.85 (1.52)
Statistical Analysis 1: Comparison: Rituximab vs No Rituximab; T-test of the natural logarithmic transformed data; Test type: Superiority; p = 0.18, t-test, 2 sided; Using Natural Log Transformed Data

2. Secondary Outcome: Maximum of the Urine Protein/Creatinine Ratio Observed Between Post-Transplant Months 3-12
Description: Maximum of the Urine Protein/Creatinine Ratio Observed Between Post-Transplant Months 3-12 will be compared between the two treatment arms using an intent-to-treat approach.
Time Frame: Post-Transplant Months 3-12
Population: Intent-to-Treat Analysis
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | Rituximab | No Rituximab
Number analyzed (Participants) | 15 | 15
ratio | 0.50 (1.53) | 0.35 (1.34)
Statistical Analysis 1: Comparison: Rituximab vs No Rituximab; T-test of Natural Log Transformed Data; Test type: Superiority; p = 0.49, t-test, 2 sided

3. Secondary Outcome: Renal Function as Measured by eGFR (Estimated Glomerular Filtration Rate)
Description: Renal function as measured by eGFR (estimated glomerular filtration rate) using the MDRD formula
Time Frame: 12 months post-transplant
Population: Intent-to-Treat Analysis
Measure: Mean (Standard Error); unit: ml/min/1.73 m^2
Arm/Group | Rituximab | No Rituximab
Number analyzed (Participants) | 15 | 15
ml/min/1.73 m^2 | 57.1 (8.4) | 66.9 (6.6)
Statistical Analysis 1: Comparison: Rituximab vs No Rituximab; T-test; Test type: Superiority; p = 0.37, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rituximab | No Rituximab
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=15) | No Rituximab (N=15)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pneumonia
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pulmonary Edema
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=15) | No Rituximab (N=15)
Abnormal GGT (Investigations) | 1 | 1
Acute Anemia (Blood and lymphatic system disorders) | 1 | 1
Acute T Cell Mediated Rejection (Immune system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 3
Ascites (Hepatobiliary disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bilateral Carpal Tunnel (Nervous system disorders) | 0 | 1
BK Virus Replication (Infections and infestations) | 3 | 0
Bladder Spasm (Renal and urinary disorders) | 1 | 1
C-Diff Infection (Infections and infestations) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Decrease Vision (Eye disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Elevated Creatinine (Investigations) | 3 | 6
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0
Evacuation of Subcapsular Hematoma (Blood and lymphatic system disorders) | 1 | 0
Flu Like Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Fluid Overload (Metabolism and nutrition disorders) | 2 | 0
Gastrointestinal Upset (Gastrointestinal disorders) | 1 | 0
Generalized Body Pain (General disorders) | 0 | 1
Generalized Edema (Metabolism and nutrition disorders) | 0 | 1
Scrotal Edema (Metabolism and nutrition disorders) | 0 | 1
Edema Extremeties (Metabolism and nutrition disorders) | 1 | 0
Bilateral Lower Extremities Edema (Metabolism and nutrition disorders) | 0 | 1
Legs Edema (Metabolism and nutrition disorders) | 0 | 1
Acute Tubular Necrosis (Renal and urinary disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hematuria (Vascular disorders) | 0 | 1
Hemorrhoids (Vascular disorders) | 1 | 0
Hypercoagulability (Blood and lymphatic system disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 6
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 2
Mouth Ulcers (Gastrointestinal disorders) | 1 | 0
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Nausea and Vomiting (Gastrointestinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 8
Pain at Incision Site Radiating to Scrotal Area (Injury, poisoning and procedural complications) | 1 | 0
Phimosis (Reproductive system and breast disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Post Surgical Pain (Injury, poisoning and procedural complications) | 3 | 2
Proteinuria (Renal and urinary disorders) | 3 | 4
CMV Viremia (Infections and infestations) | 2 | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Steal Syndrome (Vascular disorders) | 0 | 1
Swollen Right Lower Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Swollen Right Upper Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
T-Cell and Antibody Mediated Acute Rejection (Injury, poisoning and procedural complications) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Urinary Leak (Renal and urinary disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 7
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vaginal Yeast Infection (Infections and infestations) | 1 | 0
Viral Syndrome (Infections and infestations) | 1 | 0
Vomiting and Diarrhea (Gastrointestinal disorders) | 1 | 0
Worsening Anemia (Blood and lymphatic system disorders) | 1 | 2
Worsening Hypertension (Vascular disorders) | 2 | 4
Worsening Hyperglycemia (Endocrine disorders) | 0 | 1
Wound Infection (Injury, poisoning and procedural complications) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No